CLINICAL TRIAL: NCT06179342
Title: Comparison of New Methods of Multiple Breath Washout and Diffusion Capacity Determination (Ndd Medizintechnik Zurich, Trueflow™/Truecheck™) With Established Methods of Lung Function Diagnostics in Patients With Idiopathic Pulmonary Fibrosis, Chronic Obstructive Pulmonary Disease, Asthma and Cardiopulmonary Healthy Individuals
Brief Title: Multiple Breath Washout as a Method for Diagnosing Lung Diseases
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Boehringer Ingelheim (Industry); ndd Medizintechnik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: WI_20-1542_1
Record Dates: First submitted 2023-12-06; First posted 2023-12-21 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Fibrosis; COPD; Asthma
MeSH Terms: conditions — Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cardiopulmonary healthy: Patients in whom there is no evidence of cardiopulmonary dysfunction in the course of diagnostics
  Interventions: Diagnostic Test: Multiple-Breath-Washout
- Idiopathic pulmonary fibrosis: idiopathic pulmonary fibrosis (IPF), confirmed according to the guidelines
  Interventions: Diagnostic Test: Multiple-Breath-Washout
- Chronic obstructive pulmonary disease: Chronic obstructive pulmonary disease (COPD) with/without emphysema
  Interventions: Diagnostic Test: Multiple-Breath-Washout
- Asthma bronchiale
  Interventions: Diagnostic Test: Multiple-Breath-Washout

INTERVENTIONS:
Diagnostic Test: Multiple-Breath-Washout — One additional diagnostic test is performed using the Multiple-Breath-Washout technology

SUMMARY:
Comparison of the new multiple-breath washout method (ndd Medizintechnik Zürich, Trueflow™/Truecheck™) with established methods of lung function diagnostics in patients with idiopathic pulmonary fibrosis, chronic obstructive pulmonary disease, asthma and cardiopulmonary healthy individuals.

DETAILED DESCRIPTION:
This diagnostic, prospective, clinical study aims to investigate whether the lung function data measured with the EasyOnePro®LAB device correlates with the lung function data from established measurement methods used in routine clinical practice. It is to be investigated whether the EasyOnePro®LAB measurement leads to equivalent results even with a shorter measurement duration due to an improved evaluation. This is relevant for a broader clinical application in the future.

It will also be tested whether the fact that the EasyOnePro®LAB measurement can be carried out largely independently of the employee also leads to better reproducibility of the results. To this end, the intra-individual deviations in repeated measurements will be compared between the methods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* existing consent
* confirmed diagnosis of one of the following diseases
* idiopathic pulmonary fibrosis (IPF), confirmed according to the guidelines
* chronic obstructive pulmonary disease (COPD) with/without emphysema
* bronchial asthma
* or patients who are admitted with suspected cardiopulmonary dysfunction (e.g. with unclear dyspnoea) and in whom there is no evidence of cardiopulmonary dysfunction during the diagnostic process (comparison group of "healthy" patients).
* Indication for routine performance of the following pulmonary function tests during the current inpatient stay: Whole Body Plethysmography & Diffusion Capacity of the Lung (single-breath)

Exclusion Criteria:

* Age < 18 years
* Simultaneous presence of at least two of the following diseases (IPF, COPD/emphysema, asthma, pulmonary arterial hypertension)
* any medical, psychological or other condition that restricts the patient's ability to give informed consent for voluntary participation in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the study center with one of the above-mentioned diseases
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index | immediately ofter the procedure
  comparison of the lung clearance index of the different patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Lars Hagmeyer, PD Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, North Rhine-Westphalia, Germany